CLINICAL TRIAL: NCT05573412
Title: Comparison of the Proliferative Potential of Human Peripheral Blood Stem Cells Based on Demographic Factors and Cryopreservation Time
Brief Title: Comparison of Proliferative Potential of H-PBSC Based on Demographics and Cryopreservation Time
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Florida (Other)
Responsible Party: Sponsor
Other Study IDs: PBSC
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood stem cells previously preserved in cryostorage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Particpants: Group contains all participants as this is a systemic review of stem cell cryopreservation techniques
  Interventions: Other: Cellular analysis

INTERVENTIONS:
Other: Cellular analysis — Previously cryopreserved samples will be analyzed for total nucleated cell count (TNC), cell viability and proliferative potential

SUMMARY:
The goal of this observational study is to observe stored stem cells and determine their capability to grow based on several factors. The main two factors focused on in this study are as follows:

* Time stem cells have spent in cryopreservation
* Demographic factors (gender, race, age)

DETAILED DESCRIPTION:
This study is a secondary, correlational, single-center laboratory study involving the analysis of previously obtained PBSC samples at the Andrews Research & Education Foundation (AREF). Individuals who previously provided samples for a primary study that has a concluded will be reconsented for this study. No manipulation of samples will occur until Broad Informed Consent has been obtained. Upon Broad Informed Consent being granted, the samples will be removed from cryopreservation and analyzed in a laboratory setting.

Each sample's total nucleated cell count (TNC), cell viability, and proliferative potential will be analyzed. Measurements will be performed at different time intervals and the results will be recorded in a password protected system.

These parameters will be followed for each available PBSC sample regardless of time spent in cryopreservation to examine if variation in time spent under cryopreservation had an impact on overall cell viability and proliferative potential.

Following conclusion of the cell viability data acquisition stage of the study, the data will be further analyzed to determine if there are any statistically relevant correlations between various demographic factors and the viabilities of the PBSC samples. The secondary, demographic factors to be examined include the sample patient's age, sex, and race. The data analysis will determine whether these factors in addition to length of time spent under cryopreservation influenced the PBSC samples' viability and proliferative potential upon the samples being removed from cryopreservation and prepared for analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Prior primary study at Andrews Research & Education Foundation must be completed
* Additional biospecimens continue to be in a cryopreserved state at Andrews Research & Education Foundation Regenerative Medicine Center (RMC)
* Subject is willing and able to provide Broad Informed Consent for secondary study

Exclusion Criteria:

* Subjects whose biospecimens did not maintain primary study sample labels
* Subject is not willing and able to provide Broad Informed Consent for secondary study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target study population for this study is patients of any gender (age 18 or above) that has already completed a study at Andrews Research & Education Foundation and has cryopreserved blood samples at the Andrews Research & Education Foundation Regenerative Medicine Center (RMC)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-08-16 (Estimated); Study Completion 2023-08-16 (Estimated)

PRIMARY OUTCOMES:
Beckman-Coulter Flow Cytometer | At enrollment
  Machine that provides a digital view of cells that are categorized utilizing laser light to differentiate cell types while samples are suspended in a fast-flowing liquid; will be utilized to determine proliferative potential, total nucleated cell count, and cell viability of each cryopreserved sample

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anz, MD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- Andrews Research & Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gratwohl A, Hermans J, Baldomero H. Hematopoietic precursor cell transplants in Europe: activity in 1994. Report from the European Group for Blood and Marrow Transplantation (EBMT). Bone Marrow Transplant. 1996 Feb;17(2):137-48. PMID 8640158
- [Background] Korbling M, Freireich EJ. Twenty-five years of peripheral blood stem cell transplantation. Blood. 2011 Jun 16;117(24):6411-6. doi: 10.1182/blood-2010-12-322214. Epub 2011 Apr 1. PMID 21460243
- [Background] Schmitz N, Bacigalupo A, Hasenclever D, Nagler A, Gluckman E, Clark P, Bourquelot P, Greinix H, Frickhofen N, Ringden O, Zander A, Apperley JF, Gorin C, Borkett K, Schwab G, Goebel M, Russell NH, Gratwohl A. Allogeneic bone marrow transplantation vs filgrastim-mobilised peripheral blood progenitor cell transplantation in patients with early leukaemia: first results of a randomised multicentre trial of the European Group for Blood and Marrow Transplantation. Bone Marrow Transplant. 1998 May;21(10):995-1003. doi: 10.1038/sj.bmt.1701234. PMID 9632272
- [Background] Blaise D, Kuentz M, Fortanier C, Bourhis JH, Milpied N, Sutton L, Jouet JP, Attal M, Bordigoni P, Cahn JY, Boiron JM, Schuller MP, Moatti JP, Michallet M. Randomized trial of bone marrow versus lenograstim-primed blood cell allogeneic transplantation in patients with early-stage leukemia: a report from the Societe Francaise de Greffe de Moelle. J Clin Oncol. 2000 Feb;18(3):537-46. doi: 10.1200/JCO.2000.18.3.537. PMID 10653869
- [Background] Cutler C, Antin JH. Peripheral blood stem cells for allogeneic transplantation: a review. Stem Cells. 2001;19(2):108-17. doi: 10.1634/stemcells.19-2-108. PMID 11239165
- [Background] Nehrer S, Spector M, Minas T. Histologic analysis of tissue after failed cartilage repair procedures. Clin Orthop Relat Res. 1999 Aug;(365):149-62. doi: 10.1097/00003086-199908000-00020. PMID 10627699
- [Background] Mithoefer K, Williams RJ 3rd, Warren RF, Potter HG, Spock CR, Jones EC, Wickiewicz TL, Marx RG. The microfracture technique for the treatment of articular cartilage lesions in the knee. A prospective cohort study. J Bone Joint Surg Am. 2005 Sep;87(9):1911-20. doi: 10.2106/JBJS.D.02846. PMID 16140804
- [Background] Minas T, Ogura T, Bryant T. Autologous Chondrocyte Implantation. JBJS Essent Surg Tech. 2016 Jun 22;6(2):e24. doi: 10.2106/JBJS.ST.16.00018. eCollection 2016 Jun 22. PMID 30237933
- [Background] Fortier LA, Potter HG, Rickey EJ, Schnabel LV, Foo LF, Chong LR, Stokol T, Cheetham J, Nixon AJ. Concentrated bone marrow aspirate improves full-thickness cartilage repair compared with microfracture in the equine model. J Bone Joint Surg Am. 2010 Aug 18;92(10):1927-37. doi: 10.2106/JBJS.I.01284. PMID 20720135
- [Background] Lee KB, Hui JH, Song IC, Ardany L, Lee EH. Injectable mesenchymal stem cell therapy for large cartilage defects--a porcine model. Stem Cells. 2007 Nov;25(11):2964-71. doi: 10.1634/stemcells.2006-0311. Epub 2007 Jul 26. PMID 17656639
- [Background] McIlwraith CW, Frisbie DD, Rodkey WG, Kisiday JD, Werpy NM, Kawcak CE, Steadman JR. Evaluation of intra-articular mesenchymal stem cells to augment healing of microfractured chondral defects. Arthroscopy. 2011 Nov;27(11):1552-61. doi: 10.1016/j.arthro.2011.06.002. Epub 2011 Aug 20. PMID 21862278
- [Background] Nejadnik H, Hui JH, Feng Choong EP, Tai BC, Lee EH. Autologous bone marrow-derived mesenchymal stem cells versus autologous chondrocyte implantation: an observational cohort study. Am J Sports Med. 2010 Jun;38(6):1110-6. doi: 10.1177/0363546509359067. Epub 2010 Apr 14. PMID 20392971
- [Background] Tay LX, Ahmad RE, Dashtdar H, Tay KW, Masjuddin T, Ab-Rahim S, Chong PP, Selvaratnam L, Kamarul T. Treatment outcomes of alginate-embedded allogenic mesenchymal stem cells versus autologous chondrocytes for the repair of focal articular cartilage defects in a rabbit model. Am J Sports Med. 2012 Jan;40(1):83-90. doi: 10.1177/0363546511420819. Epub 2011 Sep 13. PMID 21917609
- [Background] Wakitani S, Goto T, Pineda SJ, Young RG, Mansour JM, Caplan AI, Goldberg VM. Mesenchymal cell-based repair of large, full-thickness defects of articular cartilage. J Bone Joint Surg Am. 1994 Apr;76(4):579-92. doi: 10.2106/00004623-199404000-00013. PMID 8150826
- [Background] Saw KY, Hussin P, Loke SC, Azam M, Chen HC, Tay YG, Low S, Wallin KL, Ragavanaidu K. Articular cartilage regeneration with autologous marrow aspirate and hyaluronic Acid: an experimental study in a goat model. Arthroscopy. 2009 Dec;25(12):1391-400. doi: 10.1016/j.arthro.2009.07.011. Epub 2009 Sep 17. PMID 19962065
- [Background] Saw KY, Anz A, Merican S, Tay YG, Ragavanaidu K, Jee CS, McGuire DA. Articular cartilage regeneration with autologous peripheral blood progenitor cells and hyaluronic acid after arthroscopic subchondral drilling: a report of 5 cases with histology. Arthroscopy. 2011 Apr;27(4):493-506. doi: 10.1016/j.arthro.2010.11.054. Epub 2011 Feb 19. PMID 21334844
- [Background] Saw KY, Anz A, Siew-Yoke Jee C, Merican S, Ching-Soong Ng R, Roohi SA, Ragavanaidu K. Articular cartilage regeneration with autologous peripheral blood stem cells versus hyaluronic acid: a randomized controlled trial. Arthroscopy. 2013 Apr;29(4):684-94. doi: 10.1016/j.arthro.2012.12.008. Epub 2013 Feb 4. PMID 23380230
- [Background] Saw KY, Anz AW, Ng RC, Jee CS, Low SF, Dorvault C, Johnson KB. Arthroscopic Subchondral Drilling Followed by Injection of Peripheral Blood Stem Cells and Hyaluronic Acid Showed Improved Outcome Compared to Hyaluronic Acid and Physiotherapy for Massive Knee Chondral Defects: A Randomized Controlled Trial. Arthroscopy. 2021 Aug;37(8):2502-2517. doi: 10.1016/j.arthro.2021.01.067. Epub 2021 Jul 12. PMID 34265388
- [Background] Duhrsen U, Villeval JL, Boyd J, Kannourakis G, Morstyn G, Metcalf D. Effects of recombinant human granulocyte colony-stimulating factor on hematopoietic progenitor cells in cancer patients. Blood. 1988 Dec;72(6):2074-81. PMID 3264199
- [Background] Matsunaga T, Sakamaki S, Kohgo Y, Ohi S, Hirayama Y, Niitsu Y. Recombinant human granulocyte colony-stimulating factor can mobilize sufficient amounts of peripheral blood stem cells in healthy volunteers for allogeneic transplantation. Bone Marrow Transplant. 1993 Feb;11(2):103-8. PMID 7679596
- [Background] Lane TA, Law P, Maruyama M, Young D, Burgess J, Mullen M, Mealiffe M, Terstappen LW, Hardwick A, Moubayed M, et al. Harvesting and enrichment of hematopoietic progenitor cells mobilized into the peripheral blood of normal donors by granulocyte-macrophage colony-stimulating factor (GM-CSF) or G-CSF: potential role in allogeneic marrow transplantation. Blood. 1995 Jan 1;85(1):275-82. PMID 7528570
- [Background] Skulimowska I, Sosniak J, Gonka M, Szade A, Jozkowicz A, Szade K. The biology of hematopoietic stem cells and its clinical implications. FEBS J. 2022 Dec;289(24):7740-7759. doi: 10.1111/febs.16192. Epub 2021 Sep 29. PMID 34496144
- [Background] Granick JL, Simon SI, Borjesson DL. Hematopoietic stem and progenitor cells as effectors in innate immunity. Bone Marrow Res. 2012;2012:165107. doi: 10.1155/2012/165107. Epub 2012 Jun 19. PMID 22762001
- [Background] Oh J, Lee YD, Wagers AJ. Stem cell aging: mechanisms, regulators and therapeutic opportunities. Nat Med. 2014 Aug;20(8):870-80. doi: 10.1038/nm.3651. PMID 25100532
- [Background] Ahmed AS, Sheng MH, Wasnik S, Baylink DJ, Lau KW. Effect of aging on stem cells. World J Exp Med. 2017 Feb 20;7(1):1-10. doi: 10.5493/wjem.v7.i1.1. eCollection 2017 Feb 20. PMID 28261550
- [Background] Schultz MB, Sinclair DA. When stem cells grow old: phenotypes and mechanisms of stem cell aging. Development. 2016 Jan 1;143(1):3-14. doi: 10.1242/dev.130633. PMID 26732838
- [Background] Boyette LB, Tuan RS. Adult Stem Cells and Diseases of Aging. J Clin Med. 2014 Jan 21;3(1):88-134. doi: 10.3390/jcm3010088. PMID 24757526
- [Background] Rossi DJ, Bryder D, Zahn JM, Ahlenius H, Sonu R, Wagers AJ, Weissman IL. Cell intrinsic alterations underlie hematopoietic stem cell aging. Proc Natl Acad Sci U S A. 2005 Jun 28;102(26):9194-9. doi: 10.1073/pnas.0503280102. Epub 2005 Jun 20. PMID 15967997
- [Background] Sudo K, Ema H, Morita Y, Nakauchi H. Age-associated characteristics of murine hematopoietic stem cells. J Exp Med. 2000 Nov 6;192(9):1273-80. doi: 10.1084/jem.192.9.1273. PMID 11067876
- [Background] Verovskaya E, Broekhuis MJ, Zwart E, Ritsema M, van Os R, de Haan G, Bystrykh LV. Heterogeneity of young and aged murine hematopoietic stem cells revealed by quantitative clonal analysis using cellular barcoding. Blood. 2013 Jul 25;122(4):523-32. doi: 10.1182/blood-2013-01-481135. Epub 2013 May 29. PMID 23719303
- [Background] Morrison SJ, Wandycz AM, Akashi K, Globerson A, Weissman IL. The aging of hematopoietic stem cells. Nat Med. 1996 Sep;2(9):1011-6. doi: 10.1038/nm0996-1011. PMID 8782459
- [Background] Geiger H, True JM, de Haan G, Van Zant G. Age- and stage-specific regulation patterns in the hematopoietic stem cell hierarchy. Blood. 2001 Nov 15;98(10):2966-72. doi: 10.1182/blood.v98.10.2966. PMID 11698278
- [Background] Chakkalakal JV, Jones KM, Basson MA, Brack AS. The aged niche disrupts muscle stem cell quiescence. Nature. 2012 Oct 18;490(7420):355-60. doi: 10.1038/nature11438. Epub 2012 Sep 26. PMID 23023126
- [Background] Araujo AB, Salton GD, Angeli MH, Furlan JM, Schmalfuss T, Rohsig LM. Effects of cell concentration, time of fresh storage, and cryopreservation on peripheral blood stem cells: PBSC fresh storage and cryopreservation. Transfus Apher Sci. 2022 Feb;61(1):103298. doi: 10.1016/j.transci.2021.103298. Epub 2021 Oct 21. PMID 34696981
- [Background] Hsu JW, Farhadfar N, Murthy H, Logan BR, Bo-Subait S, Frey N, Goldstein SC, Horowitz MM, Lazarus H, Schwanke JD, Shah NN, Spellman SR, Switzer GE, Devine SM, Shaw BE, Wingard JR. The Effect of Donor Graft Cryopreservation on Allogeneic Hematopoietic Cell Transplantation Outcomes: A Center for International Blood and Marrow Transplant Research Analysis. Implications during the COVID-19 Pandemic. Transplant Cell Ther. 2021 Jun;27(6):507-516. doi: 10.1016/j.jtct.2021.03.015. Epub 2021 Mar 22. PMID 33865804
- [Background] Underwood J, Rahim M, West C, Britton R, Skipworth E, Graves V, Sexton S, Harris H, Schwering D, Sinn A, Pollok KE, Robertson KA, Goebel WS, Hege KM. How old is too old? In vivo engraftment of human peripheral blood stem cells cryopreserved for up to 18 years - implications for clinical transplantation and stability programs. World J Stem Cells. 2020 May 26;12(5):359-367. doi: 10.4252/wjsc.v12.i5.359. PMID 32547684
- [Background] Pavlu J, Auner HW, Szydlo RM, Sevillano B, Palani R, O'Boyle F, Chaidos A, Jakob C, Kanfer E, MacDonald D, Milojkovic D, Rahemtulla A, Bradshaw A, Olavarria E, Apperley JF, Pello OM. Analysis of hematopoietic recovery after autologous transplantation as method of quality control for long-term progenitor cell cryopreservation. Bone Marrow Transplant. 2017 Dec;52(12):1599-1601. doi: 10.1038/bmt.2017.113. Epub 2017 Jun 26. PMID 28650454
- [Background] Liseth K, Ersvaer E, Abrahamsen JF, Nesthus I, Ryningen A, Bruserud O. Long-term cryopreservation of autologous stem cell grafts: a clinical and experimental study of hematopoietic and immunocompetent cells. Transfusion. 2009 Aug;49(8):1709-19. doi: 10.1111/j.1537-2995.2009.02180.x. PMID 19392777